CLINICAL TRIAL: NCT05938244
Title: Cardiac and Pulmonary Assessment in Egyptian Patients With Rheumatoid Arthritis and Their Correlation With Disease Activity
Brief Title: Cardiac and Pulmonary Assessment in Egyptian Patients With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yosra Yousif Mahmoud nasser, Resident doctor, Assiut University
Other Study IDs: Cardiopulmonary RA
Record Dates: First submitted 2023-06-25; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Rheumatoid Arthritis
Keywords: cardiac pulmonary rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case/ diseased patients: ultra sound anterior chest wall echocardiogram pulmonary function test diaphragmatic ultra sound lipid profile Rheumatoid factor Anti-ccp
- control/ normal population: ultra sound anterior chest wall echocardiogram pulmonary function test diaphragmatic ultra sound lipid profile Rheumatoid factor Anti-ccp

SUMMARY:
To determine cardiac and pulmonary involvement in RA patients To assess the correlation between cardiopulmonary findings in RA patients with disease activity.

To compare between diaphragmatic ultrasonography and PFT i.e. spirometry as a screening tool for restrictive pulmonary disorders.

To assess correlation between anterior chest wall ultrasound and pulmonary function test in RA patients.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inﬂammatory autoimmune disease with systemic manifestations targeting primarily synovial joints and periarticular tissues, with a 1-3% prevalence, it is the most prevalent form of inflammatory arthritis.(1,2) Although synovitis is the pathological hallmark of RA, numerous extra-articular symptoms and comorbidities are probably present.(3) Cardiovascular and pulmonary system diseases are the two main causes of death in RA patients, and their symptoms are the most serious.(2,3) Patients with RA have a 50% greater risk of CV mortality and a two-fold increased risk of myocardial infarction, which is the most common cause of death in this population. (4) Echocardiographic examination is considered a good predictive tool for some cardiac conditions with early findings while no clinical signs is yet found on these patients. (5) The second major cause of death in patients with RA is respiratory disease, which occurs in 30-40% of patients.(6) Sometimes the disease is silent until it has lung complications, which come before joint problems. RA may affect the lung interstitium, airways, and pleurae, while pulmonary vascular involvement is less frequent.(7) Diaphragmatic ultrasound can be used to determine the prevalence of interstitial lung disease involvement in RA as a restrictive disorder. The association between pulmonary function tests (PFTs), potential risk factors, and clinical correlation must be calculated.(8)(9) Anterior chest wall (ACW ) joints undergo joint changes and can be involved along the course of RA yet seems to be underestimated(1) Ultrasonography of ACW can detect those changes even before being clinically evident (10)

ELIGIBILITY:
Inclusion Criteria:

* Any patient satisfying 2010 ACR/ EULAR RA classification criteria

Exclusion Criteria:

* Patients with definite diagnosis for any other systemic autoimmune disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all Egyptian patients admitted to Assuit university hospitals with rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
To determine cardiac and pulmonary involvement in RA patients | 1 year
  By using spirometry, echocardiography

SECONDARY OUTCOMES:
To assess the correlation between cardiopulmonary findings in RA patients with disease activity | 1 year
  Using DAS28 as a measurement tool for activity
To compare between diaphragmatic ultrasonography and PFT i.e. spirometry as a screening tool for restrictive pulmonary disorders | 1 year
  Using diaphragmatic ultrasonography and pulmonary function test
To assess correlation between anterior chest wall ultrasound and pulmonary function test in RA patients | 1 year
  Anterior chest wall musculoskeletal ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Sara F. Ahmed, Lecturer, Study Chair — Assiut University; Manal M. Hassanien, Assistent prof., Study Chair — Assiut University; Samar H. Goma, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Henriquez P, Solano C, Pena A, Leon-Hernandez S, Hernandez-Diaz C, Gutierrez M, Pineda C. Sternoclavicular joint involvement in rheumatoid arthritis: clinical and ultrasound findings of a neglected joint. Arthritis Care Res (Hoboken). 2013 Jul;65(7):1177-82. doi: 10.1002/acr.21958. PMID 23335586
- [Background] Hannawi SM, Hannawi H, Al Salmi I. Cardiovascular Risk in Rheumatoid Arthritis: Literature Review. Oman Med J. 2021 May 31;36(3):e262. doi: 10.5001/omj.2021.25. eCollection 2021 May. PMID 34164156
- [Background] Figus FA, Piga M, Azzolin I, McConnell R, Iagnocco A. Rheumatoid arthritis: Extra-articular manifestations and comorbidities. Autoimmun Rev. 2021 Apr;20(4):102776. doi: 10.1016/j.autrev.2021.102776. Epub 2021 Feb 17. PMID 33609792
- [Background] Choy E, Ganeshalingam K, Semb AG, Szekanecz Z, Nurmohamed M. Cardiovascular risk in rheumatoid arthritis: recent advances in the understanding of the pivotal role of inflammation, risk predictors and the impact of treatment. Rheumatology (Oxford). 2014 Dec;53(12):2143-54. doi: 10.1093/rheumatology/keu224. Epub 2014 Jun 6. PMID 24907149
- [Background] Tekeli̇ AH. Pulmonary and cardiac involvement in patients with rheumatoid arthritis and ankylosing spondylitis. Eur Res J. 2023 Jan 14;1-10.
- [Background] Pinheiro FA, Souza DC, Sato EI. A Study of Multiple Causes of Death in Rheumatoid Arthritis. J Rheumatol. 2015 Dec;42(12):2221-8. doi: 10.3899/jrheum.150166. Epub 2015 Oct 15. PMID 26472415
- [Background] Alunno A, Gerli R, Giacomelli R, Carubbi F. Clinical, Epidemiological, and Histopathological Features of Respiratory Involvement in Rheumatoid Arthritis. Biomed Res Int. 2017;2017:7915340. doi: 10.1155/2017/7915340. Epub 2017 Nov 7. PMID 29238722
- [Background] Salaffi F, Carotti M, Di Carlo M, Tardella M, Giovagnoni A. High-resolution computed tomography of the lung in patients with rheumatoid arthritis: Prevalence of interstitial lung disease involvement and determinants of abnormalities. Medicine (Baltimore). 2019 Sep;98(38):e17088. doi: 10.1097/MD.0000000000017088. PMID 31567944
- [Background] Kelly C, Iqbal K, Iman-Gutierrez L, Evans P, Manchegowda K. Lung involvement in inflammatory rheumatic diseases. Best Pract Res Clin Rheumatol. 2016 Oct;30(5):870-888. doi: 10.1016/j.berh.2016.10.004. Epub 2016 Nov 9. PMID 27964793
- [Background] Mortada MA, Abdelrahman FI, Abdul-Sattar A, Mansour W. Relation between pulmonary function tests and ultrasonographic changes of asymptomatic anterior chest wall joints in rheumatoid arthritis patients. Egypt J Bronchol. 2022 Dec;16(1):8.